CLINICAL TRIAL: NCT00354211
Title: TREASURE: Treatment With Minimally-Invasive Cardiac Output for Assessment of User Derived Results Evaluating Economic Benefit
Brief Title: Using Minimally Invasive Cardiac Output Data vs. Standard Care for Patients Emergently Admitted to the Intensive Care Unit Who Are Hemodynamically Unstable
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Study # 2005-06, Revision B
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Output, High; Cardiac Output, Low
Keywords: Cardiac Output; Hemodynamic Phenomena
MeSH Terms: conditions — Cardiac Output, High; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: FLOTRAC™ SYSTEM
  Interventions: Device: minimally invasive cardiac output system consisting of arterial line sensor and cardiac output bedside monitor (device)
- 2: Control Group

INTERVENTIONS:
Device: minimally invasive cardiac output system consisting of arterial line sensor and cardiac output bedside monitor (device)
  Groups: 1

SUMMARY:
The purpose of this study is to evaluate if the continuous availability of minimally invasive cardiac output data during treatment in the intensive care unit (ICU) for hemodynamic instability, in comparison to standard of care will shorten the time needed to stabilize the patient.

The researchers hypothesize that early detection of instability improves the prognosis and treatment outcome of emergency intensive care patients with hemodynamic instability.

DETAILED DESCRIPTION:
Hemodynamic instability during the first 24-hours of Intensive Care Unit (ICU) admission is associated with increased risk of subsequent morbidity and mortality. Goal-directed hemodynamic support has been successfully used in a variety of patients to improve outcome. In contrast, a similar therapeutic approach applied later, or in patients with established multi-organ failure, has no beneficial effect and may even worsen the outcome.

It is conceivable that there is a window of opportunity during the phases of hemodynamic instability where therapeutic interventions have the greatest potential to influence the subsequent course of critical illness. Large scale uses of therapeutic protocols for early intervention have been hampered by logistic problems. The burden of installing invasive hemodynamic monitoring and protocols is labor intensive and requires a continuous presence of personnel with a thorough understanding of complex physiology. Various techniques have been introduced for monitoring cardiac output, stroke volume, or their surrogates. The disadvantage of these technologies so far have included user dependence of measurements results, need for calibration, and limitations in applicability. Edwards Lifesciences has developed a new algorithm for the determination of cardiac output using arterial pressure data. The FloTrac™ system, which includes the FloTrac™ sensor and Vigileo™ monitor, is utilized to capture the arterial pressure-based cardiac output measurement, which will be hereinafter referred to as APCO (Arterial Pressure Cardiac Output). This system uses an existing arterial catheter (placed in the femoral or radial artery) and does not require calibration by an external reference method. We hypothesize that using the FloTrac™ system to continuously monitor cardiac output, in addition to traditional vital signs, cardiovascular instability will be identified earlier and result in earlier intervention. In addition, following earlier diagnosis, more precise intervention will be available. If this can be achieved, patients will likely show better outcomes by reduced length of hospital stay, ICU time, Mechanical Ventilation time, incidence of renal compromise, and other related morbidity/mortality and need less ICUresources.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly admitted to the ICU due to an emergency unplanned admission.
* Patient diagnosed with hemodynamic instability at or becomes unstable within 6 hours of ICU admission.
* Patient must require an indwelling radial or a femoral artery catheter.
* Patient is included in the study according to the specific regulations of the participating center: this may include a deferred consent, consent by designee, consent by independent physician or a combination thereof.
* Patient must be 18 years old or older.

Exclusion Criteria:

* Patients with contraindications for the placement of radial, femoral, dorsalis pedis, or other arterial cannula.
* Patients with a pulmonary artery catheter.
* Patients who are hemodynamically stable.
* Patients with history or clinical findings of aortic valve regurgitation.
* Patients being treated with an intra-aortic balloon pump.
* Female patient is pregnant.
* Patient is currently participating in an investigational drug or another device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients emergently admitted to the Intensive Care Unit who develop hemodynamic instability within 6 hours of admission.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Takala, M.D., Ph.D., Principal Investigator — University Hospital Bern (Inselspital)
Locations (3):
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere Unversity Hospital, Tampere
- University Hospital Bern (Inselspital), Bern, Switzerland

REFERENCES:
- [Result] Takala J, Ruokonen E, Tenhunen JJ, Parviainen I, Jakob SM. Early non-invasive cardiac output monitoring in hemodynamically unstable intensive care patients: a multi-center randomized controlled trial. Crit Care. 2011 Jun 15;15(3):R148. doi: 10.1186/cc10273. PMID 21676229